CLINICAL TRIAL: NCT05229861
Title: The Influence of High-Intensity Interval Training Compared to Moderate Continuous Training on Cardiorespiratory Fitness, Symptom Improvement, and Disease-specific Biomarkers in Primary Progressive Multiple Sclerosis
Brief Title: The Influence of HIIT Versus MCT on Cardiorespiratory Fitness in PPMS
Acronym: CYPRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinik Valens (Other)
Collaborators: Technische Universität Dortmund, Germany (Unknown)
Responsible Party: Principal Investigator, Jens Bansi, Dr. Jens Bansi, Head of Research & Development, Klinik Valens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CYPRO
Record Dates: First submitted 2022-01-14; First posted 2022-02-08 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Primary Progressive Multiple Sclerosis; Exercise; Cardiorespiratory Fitness
Keywords: Multiple Sclerosis; Primary Progressive Multiple Sclerosis; Exercise; High-intensity Interval Exercise; Rehabilitation; Cardiorespiratory Fitness; Cognition; Mobility limitation; Quality of Life; Fatigue; Depression; Immune signalling; Inflammation; Kynurenine pathway
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Motor Activity; Multiple Sclerosis; Mobility Limitation; Fatigue; Depression; Inflammation

STUDY DESIGN:
Intervention Model Description: Single-centre Randomized Controlled Trial (RCT)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of the principal investigator and research assistant towards group allocation is ensured by a unique subject identification code given to each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity Interval Training (HIIT) (Experimental): Participants will complete seven HR-controlled HIIT sessions within their 3-week inpatient stay, corresponding to 3 exercise bouts per week.
  Interventions: Behavioral: HIIT
- Moderate Continuous Training (MCT) (Active Comparator): MCT represents the standard treatment at Valens rehabilitation clinic. Participants will complete seven HR-controlled MCT sessions within their 3-week inpatient stay, corresponding to 3 exercise bouts per week.
  Interventions: Behavioral: MCT

INTERVENTIONS:
Behavioral: HIIT — Exercise intensity will be regulated and heart rate controlled based on the achieved maximum heart rate (HRmax) assessed during the initial Cardiopulmonary Exercise Testing. Participants will perform five high-intensity intervals (95% HRpeak) at high pedalling rates of 80-100 rpm for 90 seconds each. Intervals are interspersed by active breaks of unloaded pedalling (20W, 60-70rpm) aimed to return to 60% HRpeak (approximately 1-1.5 min). The duration of a HIIT sessions is approximately 25 minutes.
  Arms: High-intensity Interval Training (HIIT)
Behavioral: MCT — Exercise intensity will be regulated and heart rate controlled based on the achieved maximum heart rate (HRmax) assessed during the initial Cardiopulmonary Exercise Testing. Participants perform continuous bicycle ergometry at moderate intensity (60% HRpeak) and 60-70 rpm for the duration of 30 minutes.
  Arms: Moderate Continuous Training (MCT)

SUMMARY:
Endurance training revealed to be an effective means to increase cardiorespiratory fitness in persons with Multiple Sclerosis (MS), considered relevant to health-related quality of life in this population. Moreover, endurance training improves MS-related symptoms, such as reduced walking capacity, fatigue, depression, and cognitive impairment. Owing to these benefits, endurance training has evolved as an integral part of MS rehabilitation, anchored in current treatment guidelines.

In recent years, High-Intensity Interval training (HIIT) evolved as a time-efficient and safe alternative to standard care in MS rehabilitation that is Moderate Continuous Training (MCT). Indeed, HIIT has already been proven superior to MCT in improving cardiorespiratory fitness, MS-related symptoms (e.g. cognitive impairment) and, beyond, seems to elicit disease-modifying effects on MS-pathophysiology (i.e. alleviated neuroinflammation and neurodegeneration).

However, current evidence is restricted to clinical trials that include samples with mixed MS disease courses, in which persons with primary progressive MS (PPMS) are underrepresented due to comparatively low prevalence rates.

Distinct pathophysiological mechanisms and symptom constellations prohibit the generalisation of previous findings to persons with PPMS. In this population, however, evidence-based rehabilitative strategies are urgently needed, as disability progression in PPMS is poorly responsive to pharmacotherapy.

This study, aims to validate previous findings on the superior effect of HIIT compared to MCT on improving cardiorespiratory fitness, MS-related symptoms and MS pathophysiology in persons with PPMS, contributing to the development of specific recommendations to maximize the effects of exercise as a potent non-pharmacological treatment adjuvant.

ELIGIBILITY:
Inclusion Criteria:

* adult age (≥ 18 years)
* definite MS diagnosis according the 2017 revised McDonald criteria
* disease course: PPMS according to the 2013 revised Lublin criteria
* disease severity: Expanded Disability Status Scale (EDSS) score ≤ 6.0
* Informed Consent as documented by signature of participants and PI

Exclusion Criteria:

* Persons suffering from severe lower extremity spasticity or severe concomitant ´ disease states (i.e., orthopaedic, cardiovascular, metabolic, psychiatric (e.g., substance abuse), other neurological, other serious medical conditions) impairing their ability to participate.
* Persons regularly performing HIIT (2-3 times per week)
* Inability to follow the procedures of the study due to language problems (i.e., participant not fluent in oral and written German language)
* Changes in disease-modifying drugs (≤ 6 weeks)
* Immunosuppressive therapy (i.e., corticosteroids) (≤ 4 weeks)
* Stem cell treatment (≤ 6 months)
* Pregnant or breast-feeding women
* Intention to become pregnant during the course of the study
* Suspected non-compliance
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees, and other dependent persons
* occurrence of severe pulmonary or cardiovascular decompensations (i.e., blood pressure (Riva Rocci) > 240/120, HR ≥ HRmax (220-years of age) (e.g. due to renal failure, hepatic dysfunction, cardiovascular disease)
* abnormalities in electrocardiography (ECG), pulse oximetry, or spirometry during initial CPET

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness (peak oxygen consumption, VO2peak) | Three weeks (day 0 to day 21)
  Cardiorespiratory fitness will be measured by peak oxygen consumption achieved in the cardiopulmonary exercise test (CPET). Higher values indicate better cardiorespiratory fitness.

SECONDARY OUTCOMES:
Peak power output (PPO) | Three weeks (day 0 to day 21)
  PPO is assessed during CPET and represents the maximum wattage achieved until exhaustion. Higher values reflect higher PPO.
Cognitive performance | Three weeks (day 0 to day 21)
  Cognitive performance is assessed with the Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS). This test battery involves three tests to assess the main cognitive domains vulnerable to MS: information processing speed, verbal and visual memory. The battery includes the Symbol Digit modalities Test (SDMT), Californian Verbal Learning Test-II (CVLT-II) and the Brief Visuospatial Memory Test revised (BVMT-R). Processing speed is the most relevant test and is assessed by the SDMT where the patients have 90s to voice numbers as rapidly as possible that were associated with target symbols within a grid printed at the top of a Stimulus page. The final score is the correct number of substitutions in 90 s, and scores ranges between 0 and 110. Higher scores indicating better cognition.
Cognitive impairment at baseline | Baseline (day 0)
  Screening of cognitive impairment is performed using the Montreal Cognitive Assessment (MoCA). The MoCA is a 30-point paper-pencil test that can be easily completed within 10 minutes. Items of the MoCA query short-term memory recall, visuospatial abilities, executive functions, attention, concentration, working memory, language, and orientation to time and place, all of which are summed up to a total score. A MoCa total score of < 26 is a sensitive measure of cognitive impairment in otherwise healthy subjects and in persons with MS.
Walking capacity | Three weeks (day 0 to day 21)
  Walking capacity is assessed via the six-minute walk test (6-MWT). The 6-MWT is used to determine the total distance in meters covered within six minutes when walking back and forth on a 30 metres hallway, as a measure of endurance walking capacity. Longer distance covered in metres reflects higher walking capacity.
Physical and psychological Impairment | Three weeks (day 0 to day 21)
  Physical and psychological Impairment is queried using the Multiple Sclerosis Impact Scale-29 (MSIS-29).The MSIS-29 contains a total of 29 items, split into two subscales, that adress physical impairment (20 items) and psychological impairment (9 items). Each item is ranked on a 5-point Likert scale with higher scores indicating higher physical and psychological impairment.
Fatigue | Three weeks (day 0 to day 21)
  Fatigue is assessed by means of the Fatigue Motor and Cognitive Scale (FSMC), that allows separate rating of motor and cognitive fatigue, based on a 5-point Likert scale (range 1-5). Scores range from 20-100 for the total, and from 10-50 for each subscale. Higher scores indicate a higher level of fatigue.
Anxiety and depressive symptoms | Three weeks (day 0 to day 21)
  Anxiety and depressive symptoms are assessed with the Hospital Anxiety and Depression Scale (HADS). The HADS was created as a 14-item scale for adults with physical ailments. On a 4-point Likert scale (range 0-3), patients rate anxiety (7 items) and depressive symptoms (7 items), respectively. Higher scores indicate a higher level of anxiety or depressive symptoms.
Kynurenine pathway (KP) metabolites | Three weeks (day 0 to day 21)
  Changes in KP metabolites are assessed to investigate the biological mechanisms that may underpin clinical improvement in persons with PPMS. The KP is dysregulated in persons with MS and is sensitive to exercise-related changes.
  KP metabolites include tryptophan, kynurenine, kynurenic acid, quinolinic acid, indolamine 2,3-dioxygenase, and tryptophan 2,3-dioxygenase. Higher levels of kynurenic acid and tryptophan, and lower levels of kynurenine, kynurenic acid, quinolinic acid, indolamine 2,3-dioxygenase, and tryptophan 2,3-dioxygenase indicate a beneficial effect of KP regulation.
  KP metabolites are analyzed via targeted metabolomics (HPLC MS/MS).
Immune status (blood cells) | Time Frame: Three weeks (day 0 to day 21)
  Numbers and proportions of circulating immune cells associated with MS and exercise (Th17 cell, cytotoxic T-cells, naïve T-cells, memory T-cells, NK-cells, Monocytes) are assessed, with higher values indicating higher levels of inflammation. Number and proportion of circulating regulatory T cells with higher values indicating lower levels of inflammation.
  Numbers of proportions of these circulating immune cells are determined by flow cytometric characterization of Th17 cell, cytotoxic T-cells, naïve T-cells, memory T-cells, NK-cells, and Monocytes.
Immune status (pro-inflammatory cytokines) | Time Frame: Three weeks (day 0 to day 21)
  The pro-inflammatory cytokines IL-6, IFN-γ, TNF-α are known to be produced or secreted in response to chronic exercise and modify immune homeostasis. Higher values indicate higher levels of inflammation.
  Serum concentrations of IL-6, IFN-γ, and TNF-α are determined using commercial enzyme-linked immunosorbent assays (ELISAs) according to the manufacturer's instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Gonzenbach, MD, Study Director — Klinik Valens; Bansi Jens, PhD, Principal Investigator — Klinik Valens
Locations (1):
- Klinik Valens, Valens rehabilitation clinic, Valens, Canton of St. Gallen, Switzerland

REFERENCES:
- [Result] Bansi J, Koliamitra C, Bloch W, Joisten N, Schenk A, Watson M, Kool J, Langdon D, Dalgas U, Kesselring J, Zimmer P. Persons with secondary progressive and relapsing remitting multiple sclerosis reveal different responses of tryptophan metabolism to acute endurance exercise and training. J Neuroimmunol. 2018 Jan 15;314:101-105. doi: 10.1016/j.jneuroim.2017.12.001. Epub 2017 Dec 6. PMID 29224960
- [Result] Zimmer P, Bloch W, Schenk A, Oberste M, Riedel S, Kool J, Langdon D, Dalgas U, Kesselring J, Bansi J. High-intensity interval exercise improves cognitive performance and reduces matrix metalloproteinases-2 serum levels in persons with multiple sclerosis: A randomized controlled trial. Mult Scler. 2018 Oct;24(12):1635-1644. doi: 10.1177/1352458517728342. Epub 2017 Aug 21. PMID 28825348
- [Result] Joisten N, Proschinger S, Rademacher A, Schenk A, Bloch W, Warnke C, Gonzenbach R, Kool J, Bansi J, Zimmer P. High-intensity interval training reduces neutrophil-to-lymphocyte ratio in persons with multiple sclerosis during inpatient rehabilitation. Mult Scler. 2021 Jun;27(7):1136-1139. doi: 10.1177/1352458520951382. Epub 2020 Sep 3. PMID 32880214
- [Result] Joisten N, Rademacher A, Warnke C, Proschinger S, Schenk A, Walzik D, Knoop A, Thevis M, Steffen F, Bittner S, Gonzenbach R, Kool J, Bloch W, Bansi J, Zimmer P. Exercise Diminishes Plasma Neurofilament Light Chain and Reroutes the Kynurenine Pathway in Multiple Sclerosis. Neurol Neuroimmunol Neuroinflamm. 2021 Mar 29;8(3):e982. doi: 10.1212/NXI.0000000000000982. Print 2021 May. PMID 33782190
- [Result] Lea Schlagheck M, Wucherer A, Rademacher A, Joisten N, Proschinger S, Walzik D, Bloch W, Kool J, Gonzenbach R, Bansi J, Zimmer P. VO2peak Response Heterogeneity in Persons with Multiple Sclerosis: To HIIT or Not to HIIT? Int J Sports Med. 2021 Dec;42(14):1319-1328. doi: 10.1055/a-1481-8639. Epub 2021 Jul 1. PMID 34198345
- [Result] Rademacher A, Joisten N, Proschinger S, Hebchen J, Schlagheck ML, Bloch W, Gonzenbach R, Kool J, Bansi J, Zimmer P. Do baseline cognitive status, participant specific characteristics and EDSS impact changes of cognitive performance following aerobic exercise intervention in multiple sclerosis? Mult Scler Relat Disord. 2021 Jun;51:102905. doi: 10.1016/j.msard.2021.102905. Epub 2021 Mar 18. PMID 33836459
- [Result] Rademacher A, Joisten N, Proschinger S, Bloch W, Gonzenbach R, Kool J, Langdon D, Bansi J, Zimmer P. Cognitive Impairment Impacts Exercise Effects on Cognition in Multiple Sclerosis. Front Neurol. 2021 Jan 28;11:619500. doi: 10.3389/fneur.2020.619500. eCollection 2020. PMID 33633658
- [Derived] Kupjetz M, Joisten N, Rademacher A, Gonzenbach R, Bansi J, Zimmer P. Cycling in primary progressive multiple sclerosis (CYPRO): study protocol for a randomized controlled superiority trial evaluating the effects of high-intensity interval training in persons with primary progressive multiple sclerosis. BMC Neurol. 2023 Apr 22;23(1):162. doi: 10.1186/s12883-023-03187-6. PMID 37087424